CLINICAL TRIAL: NCT00082615
Title: Neurophysiological Markers in Patients With Craniofacial Dystonia and Their Relatives
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040188; 04-N-0188
Record Dates: First submitted 2004-05-13; First posted 2004-05-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-04-21

CONDITIONS: Dystonia
Keywords: Movement Disorders; Recovery Cycle; Blink Reflex; Cervical Dystonia; Blepharospasm; Dystonia; Craniofacial Dystonia; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonia; Movement Disorders; Torticollis; Blepharospasm

SUMMARY:
This study will use a technique called blink reflex to study and compare how the brain controls muscle movement in patients with craniofacial dystonia, their first-degree relatives, and healthy, normal volunteers. People with dystonia have sustained muscle contractions that cause twisting and repetitive movements or abnormal postures. In focal dystonia, this happens in one area of the body, such as the hand, neck, or face.

Three groups of people may be eligible for this study: 1) patients 18 years of age and older with craniofacial dystonia; 2) first-degree relatives of patients with craniofacial dystonia; and 3) normal volunteers matched in age to the patients. Candidates are screened with physical and neurological examinations.

Participants undergo a blink reflex study. Patients with dystonia who are receiving botulinum toxin injections must stop the medication 3 months before participating in the study and must stop any other dystonia medications, such as benzodiazepines and anticholinergics, for 12 hours before the study. For the blink reflex procedure, subjects are seated in a comfortable chair with their hands placed on a pillow on their lap. Metal electrodes are taped to the forehead for delivering small electrical shocks that feel like very brief pinpricks. Subjects receive 25 to 50 electrical stimuli, some as single shocks and some in pairs. The electrical activity of muscles that respond to the stimuli is recorded with a computer. The study takes from about 1 to 2 hours.

DETAILED DESCRIPTION:
The objective of this study is to evaluate paired-pulse inhibition of the three responses of the electrically elicited blink reflex (BR) and the eye blink rate (EBR)in patients with craniofacial dystonia and their first degree relatives in order to determine whether abnormalities of inhibition can represent a marker of genetic predisposition for the development of dystonia. It is unclear why some relatives of patients with craniofacial dystonia do not develop dystonic symptoms. One possible explanation is that the development of dystonia is a two-stage process: first, loss of inhibition, which may be genetically determined, and second, exposure to an environmental trigger such as excessive repetitive movements. There is good evidence that focal dystonia is a genetically determined disorder, but the responsible gene remains undetermined. Patients, their first degree relatives and normal volunteers will undergo BR testing using validated electrophysiological tests of recovery cycle. The main outcome measure of the study is impaired inhibition in up to 50% of first degree relatives of patients with focal dystonia which would serve as biologic marker for the carrier state. A second outcome measure is the EBR. In those individuals with this genetic marker of impaired inhibition, future linkage analysis studies could be performed to identify the causative gene.

ELIGIBILITY:
* INCLUSION CRITERIA:

Three groups of subjects shall be studied: 1) patients with craniofacial dystonia, 2) first degree relatives of patients with craniofacial dystonia, 3) age matched control group. The inclusion of the group of relatives will be valuable to study, as these individuals have shared similar environment backgrounds as patients but remain free of symptoms. Patients and their relatives 18 years or older will be enrolled through the Human Motor Control Clinic, NINDS, NIH under protocol 93-N-0202: "Diagnosis and Natural History Protocol for Patients with Different Neurological Conditions". Patients with dystonia, enrolled in Protocol 85-N-0195, "Efficacy and Pathophysiology of Botulinum Toxin for Treatment of Involuntary Movement Disorders' will also be eligible for participation in the study. Diagnosis of dystonia will rely on review of medical record, history, and clinical evaluation. Age matched volunteers over 18 years-old entered into the study must be free of neurological disease as determined by a standard physical and neurological examination.

INCLUSION CRITERIA FOR VIDEOTAPING:

Patients with idiopathic BSP or Meige-Syndrome (=BSP plus oromandibular dystonia), their first degree relatives and age matched volunteers

Age18 years or older

Eye blink rate at rest more than 27 per minute (patients only)

EXCLUSION CRITERIA:

Patients, their first degree relatives and normal volunteers with any significant medical or psychiatric illness, pregnancy, history of epilepsy, concurrent use of tricyclic antidepressants, neuroleptic agents, or any other licit or illicit drug that could affect brainstem excitability will not be eligible for this study. Subjects who have a pacemaker, an implanted medication pump, metal objects inside the eye or skull (for example, after brain surgery or a shrapnel would) or any recent (less than 3 months) brain lesions will not be included in this study. Patients who have received botulinum toxin injection less than three months prior to the day of testing will also be excluded.

EXCLUSION CRITERIA FOR VIDEOTAPING:

Other disease with involuntary blinking (Hemifacial spasm, Tic disorder, Tardive Dyskinesia, Blepharitis)

Taking the following medications: antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines

Subject's objection to being videotaped while performing different activities

First degree relatives and age matched volunteers who are diagnosed with a neurological or psychiatric disease or medication that alter the blink frequency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2004-05-11; Study Completion 2008-04-21

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hallett M. Blepharospasm: recent advances. Neurology. 2002 Nov 12;59(9):1306-12. doi: 10.1212/01.wnl.0000027361.73814.0e. PMID 12434791